CLINICAL TRIAL: NCT00770770
Title: A Randomized, Double-masked, Pilot Study of the Safety and Efficacy of 0.5 µg/Day and 0.2 µg/Day Iluvien™ (Fluocinolone Acetonide Intravitreal Insert) 0.19 mg in Subjects With Macular Edema Secondary to Retinal Vein Occlusion
Brief Title: Fluocinolone Acetonide Intravitreal Inserts for Vein Occlusion in Retina
Acronym: FAVOR
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Alimera Sciences (Industry)
Responsible Party: Sponsor
Organization: ANI Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-01-08-006
Record Dates: First submitted 2008-10-09; First posted 2008-10-10 (Estimated); Results first posted 2015-05-28 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Macular Edema; Retinal Vein Occlusion
Keywords: Macular edema secondary to RVO
MeSH Terms: conditions — Macular Edema; Retinal Vein Occlusion | interventions — Fluocinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fluocinolone Acetonide 0.2 µg/day (Experimental): 0.2 µg/day
  Interventions: Drug: Fluocinolone Acetonide
- Fluocinolone Acetonide 0.5 µg/day (Experimental): 0.5 µg/day
  Interventions: Drug: Fluocinolone Acetonide

INTERVENTIONS:
Drug: Fluocinolone Acetonide — 0.2 µg/day
  Arms: Fluocinolone Acetonide 0.2 µg/day
Drug: Fluocinolone Acetonide — 0.5 µg/day
  Arms: Fluocinolone Acetonide 0.5 µg/day

SUMMARY:
This study will assess the safety and efficacy of FA Intravitreal Inserts in subjects with macular edema secondary to RVO.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of macular edema due to branch retinal vein occlusion (BRVO) or central retinal vein occlusion (CRVO)
* Central subfield thickness > 300 μm
* BCVA of ≥ 24 and ≤ 68 letters
* Males and non-pregnant females 18 years and over

Exclusion Criteria:

* Macular edema secondary to any condition other than RVO
* Presence of foveal atrophy, dense pigmentary changes or dense subfoveal exudates in the study eye
* Cystic intraretinal hemorrhage involving the fovea in the study eye that is responsible for vision loss
* Glaucoma or ocular hypertension (IOP > 21 mmHg or concurrent therapy at screening with IOP-lowering agents)
* Any prior treatment with intravitreal, subtenon, or periocular steroid or anti-VEGF therapy since the diagnosis of RVO in the study eye
* Any change in systemic steroid therapy within 3 months of screening
* History of vitrectomy in the study eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-05; Primary Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Kentucky Department of Ophthalmology, Lexington, Kentucky
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Cole Eye Institute, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Groups:
- Fluocinolone Acetonide: 0.2 µg/Day: Fluocinolone Acetonide: 0.2 µg/day
- Fluocinolone Acetonide: 0.5 µg/Day: Fluocinolone Acetonide: 0.5 µg/day
Period: Overall Study
Arm/Group | Fluocinolone Acetonide: 0.2 µg/Day | Fluocinolone Acetonide: 0.5 µg/Day
Started | 14 | 6
Completed | 4 | 5
Not Completed | 10 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Death | 0 | 1
Not completed — Study Terminated | 8 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluocinolone Acetonide 0.2 µg/Day | Fluocinolone Acetonide 0.5 µg/Day | Total
Number analyzed (Participants) | 14 | 6 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.50 (9.287) | 73.52 (13.091) | 69.30 (10.589)
Age, Customized [Number; unit: participants]
  <35 years | 0 | 0 | 0
  35-45 years | 0 | 0 | 0
  45-55 years | 2 | 0 | 2
  55-65 years | 3 | 2 | 5
  65-75 years | 6 | 0 | 6
  75-85 years | 2 | 3 | 5
  ≥85 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 7 | 2 | 9
Region of Enrollment [Number; unit: participants]
  United States | 14 | 6 | 20

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity
Description: To compare the 3 month best corrected visual acuity to baseline in subjects diagnosed with macular edema secondary to retinal vein occlusion. BCVA will be measured according to the standard procedure developed for ETDRS at 4 meters or 3 meters if the electronic (E)-ETDRS system is employed.
Time Frame: 3 months
Measure: Mean (Standard Error); unit: Letters
Arm/Group | Fluocinolone Acetonide 0.2 µg/Day | Fluocinolone Acetonide 0.5 µg/Day
Number analyzed (Participants) | 14 | 6
Letters
  Baseline | 47.0 (4.50) | 53.5 (4.13)
  Month 3 - Change from Baseline | 7.0 (2.51) | 9.2 (2.37)

ADVERSE EVENTS:
Arm/Group | Fluocinolone Acetonide: 0.2 µg/Day | Fluocinolone Acetonide: 0.5 µg/Day
Serious Adverse Events (participants affected / at risk) | 8/14 | 4/6
Other Adverse Events (participants affected / at risk) | 13/14 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluocinolone Acetonide: 0.2 µg/Day (N=14) | Fluocinolone Acetonide: 0.5 µg/Day (N=6)
Angina pectoris (Cardiac disorders) | 2 (2) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0) — #Study eye
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pseudomonas infection (Infections and infestations) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0)
Mental disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Bladder obstruction (Renal and urinary disorders) | 1 (2) | 0 (0)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cardiac pacemaker replacement (Surgical and medical procedures) | 1 (1) | 0 (0)
Cataract operation (Surgical and medical procedures) | 3 (3) | 3 (3) — #Study eye
Cataract operation (Surgical and medical procedures) | 2 (2) | 0 (0) — #Fellow eye
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluocinolone Acetonide: 0.2 µg/Day (N=14) | Fluocinolone Acetonide: 0.5 µg/Day (N=6)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Angina pectoris (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 2 (2) | 4 (4) — #Study eye
Cataract (Eye disorders) | 3 (3) | 1 (1) — #Fellow eye
Cataract subcapsular (Eye disorders) | 1 (1) | 0 (0) — #Study eye
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 1 (1) — #Study eye
Diabetic retinopathy (Eye disorders) | 1 (1) | 0 (0) — #Fellow eye
Diplopia (Eye disorders) | 1 (1) | 0 (0) — #Study eye
Diplopia (Eye disorders) | 1 (1) | 0 (0) — #Fellow eye
Dry eye (Eye disorders) | 1 (1) | 1 (1) — #Study eye
Dry eye (Eye disorders) | 1 (1) | 0 (0) — #Fellow eye
Eye irritation (Eye disorders) | 1 (1) | 0 (0) — #Study eye
Eye pain (Eye disorders) | 3 (3) | 1 (1) — #Study eye
Eye pain (Eye disorders) | 1 (1) | 0 (0) — #Fellow eye
Iris neovascularisation (Eye disorders) | 1 (1) | 0 (0) — #Study eye
Myodesopsia (Eye disorders) | 2 (2) | 1 (1) — #Study eye
Ocular hyperaemia (Eye disorders) | 2 (2) | 0 (0) — #Study eye
Optic atrophy (Eye disorders) | 1 (1) | 0 (0) — #Study eye
Optic disc haemorrhage (Eye disorders) | 0 (0) | 1 (1) — #Study eye
Optic disc vascular disorder (Eye disorders) | 1 (1) | 1 (1) — #Study eye
Papilloedema (Eye disorders) | 0 (0) | 1 (2) — #Study eye
Photophobia (Eye disorders) | 2 (2) | 0 (0) — #Study eye
Photopsia (Eye disorders) | 1 (1) | 0 (0) — #Study eye
Retinal aneurysm (Eye disorders) | 1 (1) | 0 (0) — #Fellow eye
Retinal haemorrhage (Eye disorders) | 1 (1) | 1 (1) — #Study eye
Retinal neovascularisation (Eye disorders) | 1 (1) | 0 (0) — #Study eye
Retinal oedema (Eye disorders) | 0 (0) | 1 (1) — #Study eye
Visual acuity reduced (Eye disorders) | 1 (2) | 0 (0) — #Study eye
Vitreous detachment (Eye disorders) | 1 (1) | 0 (0) — #Study eye
Vitreous detachment (Eye disorders) | 1 (1) | 0 (0) — #Fellow eye
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (4) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (3) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Sensation of foreign body (General disorders) | 2 (2) | 0 (0) — #Study eye
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pseudomonas infection (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 2 (3) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (6) | 0 (0)
Contrast media reaction (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intraocular pressure increased (Investigations) | 3 (3) | 0 (0) — #Study eye
Intraocular pressure increased (Investigations) | 1 (1) | 0 (0) — #Fellow eye
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Hemianopia (Nervous system disorders) | 1 (1) | 0 (0) — #Study eye
Hemianopia (Nervous system disorders) | 1 (1) | 0 (0) — #Fellow eye
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Bladder obstruction (Renal and urinary disorders) | 1 (3) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days